CLINICAL TRIAL: NCT00506701
Title: Pilot Study to Investigate the Effect of Tadalafil on Secondary Pulmonary Hypertension in Chronic Obstructive Pulmonary Disease
Brief Title: Effect of Tadalafil in Chronic Obstructive Lung Disease Patients Suffering From Secondary Pulmonary Hypertension
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: due to lack of finance
Sponsor: Herlev Hospital (Other)
Responsible Party: Lars C. Laursen, Herlev Hospital
Allocation: Not Applicable | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: 25
Record Dates: First submitted 2007-07-23; First posted 2007-07-25 (Estimated); Last update posted 2015-03-18 (Estimated); Status verified 2007-07

CONDITIONS: Chronic Obstructive Lung Disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Tadalafil; Phosphodiesterase 5 Inhibitors

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Tadalafil treatment 40 mg (Experimental)
  Interventions: Drug: Tadalafil

INTERVENTIONS:
Drug: Tadalafil — 40 mg tablet
  Other Names: PDE5 inhibitor

SUMMARY:
Tadalafil may lower the pulmonary artery pressure in patients with Chronic Obstructive Lung Disease and secondary pulmonary hypertension and thereby improve patients quality of life.

DETAILED DESCRIPTION:
Twenty outpatients with Chronic Obstructive Lung Disease (COPD) and secondary pulmonary hypertension are treated in a cross-over design with Tadalafil or placebo for 4 weeks. Primary effect parameter is 6 min. walking test.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Chronic obstructive lung disease

Exclusion Criteria

* Patients with asthma

Ages: 45 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2008-02; Primary Completion 2010-02 (Actual); Study Completion 2010-02 (Estimated)

PRIMARY OUTCOMES:
Change in 6 min. walking test | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Lars C Laursen, MD, Principal Investigator — University of Copenhagen
Locations (1):
- Herlev University Hospital, Herlev, Denmark